CLINICAL TRIAL: NCT01265797
Title: Cranial Electrotherapy Stimulation in the Treatment of Migraine Headaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Principal Investigator, Gretchen Tietjen, MD, Principal Investigator, University of Toledo Health Science Campus
Organization: University of Toledo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UTHSC-13
Record Dates: First submitted 2010-12-15; First posted 2010-12-23 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cranial Electrostimulator (Active Comparator): wears active cranial electrostimulation device for 20 minutes daily for 28 days
  Interventions: Device: Cranial Electrostimulator
- Sham device (Sham Comparator): wears sham device for 20 minutes daily for 28 days
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: Cranial Electrostimulator — participant wears active cranial electrostimulation device for 20 minutes daily for 28 days
  Other Names: Fisher Wallace Cranial Electrostimulator
  Arms: Cranial Electrostimulator
Device: Sham Device — participant wears sham device for 20 minutes daily for 28 days
  Arms: Sham device

SUMMARY:
Cranial electrotherapy stimulation (CES) may be a safe adjunct to medical treatment for pain relief in migraine patients. However, despite the number of CES studies done, many have been open label, single blinded, or have utilized a small group of patients.

DETAILED DESCRIPTION:
This study will evaluate the efficacy of the Fisher Wallace Cranial Stimulator in persons with chronic migraine who have not achieved satisfactory pain control on their current medications.

ELIGIBILITY:
Inclusion Criteria:

* Subjects satisfying the IHS (International Headache Society) criteria for migraine
* Subjects have not achieved satisfactory pain control on their current medication
* Ability to maintain a daily headache diary
* Stable medication use related to migraine for at least 4 weeks prior to enrollment in the study

Exclusion Criteria:

* Previous exposure to or experience with cranial electrotherapy stimulation (CES)
* Contraindications to Fisher Wallace stimulator, such as cardiac pacemakers or implantable defibrillators, known or suspected heart disease, or pregnancy
* Seizure disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-12; Primary Completion 2013-02 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Tietjen, MD, Principal Investigator — University of Toledo, HSC
Locations (1):
- University of Toledo, Health Science Campus, Toledo, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates: Dec 2010 - Jan 2013 Recruitment status: Not enrolling. Location: Neurology Clinic
Pre-assignment Details: Enrolled participants were randomized to receive verum or sham intervention. Completion of one (run-in) month headache diary was required before obtaining device.
Groups:
- Verum: Verum : wears active cranial electrostimulation device for 20 minutes daily for 28 days
- Sham: Sham: wears sham cranial electrostimulation device for 20 minutes daily for 28 days
Period: Run-in Month
Arm/Group | Verum | Sham
Started | 34 | 34
Completed | 34 | 29
Not Completed | 0 | 5
Not completed — Withdrawal by Subject | 0 | 4
Not completed — 1st seizure during run-in month | 0 | 1
Period: Blinded Month
Arm/Group | Verum | Sham
Started | 34 | 29
Completed | 24 | 27
Not Completed | 10 | 2
Not completed — Lack of Efficacy | 5 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 2 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Diary data incomplete | 0 | 1
Period: Open Label Month
Arm/Group | Verum | Sham
Started | 24 | 27
Completed | 24 | 26
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: The overall number of baseline participants used for analysis is the number completing the blinded period from the run-in period, and differs from the number of participants started in the Participant Flow Module due to drop-out and other causes listed in the participant flow module.
Groups:
- Verum: Verum : wears active Electrostimulator device daily for 20 minutes for 28 days
- Sham: Sham Device : wears Sham device daily for 20 minutes for 28 days
- Total: Total of all reporting groups
Arm/Group | Verum | Sham | Total
Number analyzed (Participants) | 24 | 27 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 27 | 51
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.67 (12.33) | 43.59 (10.25) | 43.14 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 24 | 43
  Male | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 24 | 27 | 51

OUTCOME MEASURES:

1. Primary Outcome: Mean Headache Days
Description: Mean change in headache days between 28 day run-in month and 28 day blinded month, i.e. run-in month mean minus blinded month mean. A good response is >= 50% reduction in headache days (congruent with the Guidelines for Trial of Behavioral Treatments for Recurrent Headache).
Time Frame: 28 day period during run-in month and blinded month
Measure: Mean (95% Confidence Interval); unit: headache days/ 28 day period
Arm/Group | Verum | Sham
Number analyzed (Participants) | 24 | 27
headache days/ 28 day period | 0.88 [-0.38 to 2.13] | -0.52 [-2.49 to 1.45]
Statistical Analysis 1: Comparison: Verum vs Sham; The a priori alpha level was set at p < 0.05, and a power of 0.80 (80%) was used to compute the number of subjects needed to find a meaningful difference between the verum and sham groups. Assuming that 20% of persons with the sham device and 60% of persons with CES device will meet the primary end point of ≥50% decrease in the frequency of headache days over the course of the study, 27 subjects are enrolled per group; Test type: Superiority or Other; p = 0.30, Wilcoxon (Mann-Whitney); The Mann-Whitney U test was used to compare outcome measures between two treatment groups in the run-in month minus blinded month; Mean Difference (Final Values) = 1.4

2. Secondary Outcome: Headache Days
Description: Mean change in headache days between 28 day run-in month and 28 day open label month, i.e. run-in month mean minus open label month mean. A good response is >= 50% reduction in headache days (congruent with the Guidelines for Trial of Behavioral Treatments for Recurrent Headache).
Time Frame: 28 day period in run-in month and open label month
Measure: Mean (95% Confidence Interval); unit: headache days/ 28 day period
Arm/Group | Verum | Sham
Number analyzed (Participants) | 24 | 26
headache days/ 28 day period | 0.67 [-0.63 to 1.96] | 0.76 [-1.77 to 3.22]
Statistical Analysis 1: Comparison: Verum vs Sham; Test type: Superiority or Other; p = 0.89, Wilcoxon (Mann-Whitney); The Mann-Whitney U test was used to compare secondary outcome measures between two treatment groups in the run-in month minus open label month; Mean Difference (Final Values) = -0.09

3. Secondary Outcome: Depression Score (Patient Health Questionnaire-9)
Description: Mean difference of PHQ-9 score between the run-in month and open label month, i.e. PHQ-9 score from run-in month minus open label month. The PHQ-9 is a tool for assisting in diagnosing depression (over the prior 2 week period) as well as selecting and monitoring treatment. There are nine items, with responses each ranging from 0 (not at all) to 3 (nearly every day), for a total range of 0 to 27. The higher the total the more severe the depressive symptoms.
Time Frame: 14 day recall, recorded at the end of run-in and open label months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Verum | Sham
Number analyzed (Participants) | 24 | 26
score on a scale | 1.58 [0.04 to 3.12] | 0.62 [-0.91 to 2.14]
Statistical Analysis 1: Comparison: Verum vs Sham; Test type: Superiority or Other; p = 0.30, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.96

4. Primary Outcome: Depression Score (PATIENT HEALTH QUESTIONNAIRE [PHQ] 9)
Description: Mean difference of PHQ-9 score between the run-in month and blinded month, i.e. PHQ-9 score from run-in month minus blinded month. The PHQ-9 is a tool for assisting in diagnosing depression (over the prior 2 week period) as well as selecting and monitoring treatment. There are nine items, with responses each ranging from 0 (not at all) to 3 (nearly every day), for a total range of 0 to 27. The higher the total the more severe the depressive symptoms.
Time Frame: 14 days recall; measured at end of run-in month and blinded month
Population: The number of participants included the individuals who have completed the run-in period and the blinded period. The data was analyzed 'per protocol' based on the number of participants completing the blinded period.
Measure: Mean (95% Confidence Interval); unit: depression score/14 day recall
Arm/Group | Verum | Sham
Number analyzed (Participants) | 24 | 27
depression score/14 day recall | 0 [-1.37 to 1.37] | 0.30 [-0.89 to 1.49]
Statistical Analysis 1: Comparison: Verum vs Sham; The a priori alpha level was set at p < 0.05, and beta 0.2. Assuming that 20% of persons with the sham device and 60% of persons with CES device will meet the primary end point of ≥50% decrease in the frequency of headache days over the course of the study, 27 subjects are enrolled per group. The null hypothesis: No difference in the depression score/14 day recall between the two groups; Test type: Superiority or Other; p = 0.98, Wilcoxon (Mann-Whitney); The Mann-Whitney U test was used to compare the primary and secondary outcome measures between the two treatment groups; Mean Difference (Final Values) = -0.30

5. Secondary Outcome: Headache Impact Test-6
Description: Mean difference in HIT-6 score between run-in month and blinded month. The HIT-6 is a tool for screening and monitoring change in headache disability. This disease-specific health survey is intended for adults 18 years of age and older, and is available with a standard four-week recall period. It is a 6 item questionnaire with scores for each item ranging from 6 (never) to 13 (always). The minimum overall score is 36 and the maximum is 78. Higher scores represent greater disability.
Time Frame: after run-in month, after blinded month
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Verum | Sham
Number analyzed (Participants) | 24 | 27
score on a scale | 2.13 [0.15 to 4.10] | 1.22 [-0.19 to 2.64]
Statistical Analysis 1: Comparison: Verum vs Sham; Test type: Superiority or Other; p = 0.75, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.91

6. Secondary Outcome: Headache Impact Test (HIT-6) (Measure of Disability Due to Headaches)
Description: Mean difference in HIT-6 score between run-in month and open label month. The HIT-6 is a tool for screening and monitoring change in headache disability. This disease-specific health survey is intended for adults 18 years of age and older, and is available with a standard four-week recall period. It is a 6 item questionnaire with scores for each item ranging from 6 (never) to 13 (always). The minimum overall score is 36 and the maximum is 78. Higher scores represent greater disability.
Time Frame: 28 day period in run-in month and open label month
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Verum | Sham
Number analyzed (Participants) | 24 | 26
score on a scale | 3.25 [1.39 to 5.10] | 2.65 [0.07 to 5.23]
Statistical Analysis 1: Comparison: Verum vs Sham; Test type: Superiority or Other; p = 0.73, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.6

7. Secondary Outcome: Generalized Anxiety Disorder Score (GAD 7)
Description: Mean difference in GAD 7 score between run-in month and blinded month. This is a screening tool and severity measure for generalized anxiety disorder addressing symptoms over the prior 2 weeks. It is a 7 item questionnaire with response scores for each item ranging from 0 (not at all) to 3 (every day). The range for the total score is 0 to 21, with higher scores representing greater symptoms of anxiety
Time Frame: 14 days recall; measured at end of run-in month and blinded month
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Verum | Sham
Number analyzed (Participants) | 24 | 27
score on a scale | -0.33 [-1.42 to 0.76] | 2.41 [0.51 to 4.30]
Statistical Analysis 1: Comparison: Verum vs Sham; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney) — Change in mean anxiety score/ 14 day recall from the blinded period to open label period; Mean Difference (Final Values) = -2.74

8. Secondary Outcome: Generalized Anxiety Disorder Score (GAD 7)
Description: Mean difference in GAD 7 score between run-in month and open label month. This is a screening tool and severity measure for generalized anxiety disorder addressing symptoms over the prior 2 weeks. It is a 7 item questionnaire with response scores for each item ranging from 0 (not at all) to 3 (every day). The range for the total score is 0 to 21, with higher scores representing greater symptoms of anxiety
Time Frame: 14 day recall, recorded at the end of run-in and open label months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Verum | Sham
Number analyzed (Participants) | 24 | 26
score on a scale | 1.13 [0.03 to 2.22] | 1.27 [-0.35 to 2.88]
Statistical Analysis 1: Comparison: Verum vs Sham; Test type: Superiority or Other; p = 0.98, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.14

9. Secondary Outcome: Somatic Symptom Severity (Patient Health Questionnaire 15)
Description: Mean difference in PHQ 15 score between run-in month and blinded month. The PHQ-15 comprises 15 somatic symptoms experienced over the prior 4 weeks and their severity, each symptom scored from 0 ("not bothered at all") to 2 ("bothered a lot"). The range for the overall score is between 0 and 30, with higher score representing more severe somatic symptoms
Time Frame: 28 days recall; measured at end of run-in month and blinded month
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Verum | Sham
Number analyzed (Participants) | 24 | 27
score on a scale | 0.38 [-1.29 to 2.04] | 0.33 [-0.68 to 1.34]
Statistical Analysis 1: Comparison: Verum; Test type: Superiority or Other; p = 0.97, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0.05

10. Secondary Outcome: Somatic Symptom Score (Patient Health Questionnaire-15)
Description: Mean difference in PHQ 15 score between run-in month and open label month. The PHQ-15 comprises 15 somatic symptoms experienced over the prior 4 weeks and their severity, each symptom scored from 0 ("not bothered at all") to 2 ("bothered a lot"). The range for the overall score is between 0 and 30, with higher score representing more severe somatic symptoms.
Time Frame: 28 day period in run-in month and open label month
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Verum | Sham
Number analyzed (Participants) | 24 | 26
score on a scale | 0.84 [-0.40 to 2.06] | 1.00 [-0.17 to 2.28]
Statistical Analysis 1: Comparison: Verum vs Sham; Test type: Superiority or Other; p = 0.87, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.16

11. Secondary Outcome: Epworth Sleepiness Scale Score
Description: Mean difference of Epworth Sleepiness Scale score between run-in month and blinded month. The Epworth Sleepiness Scale is used to measure excessive daytime sleepiness. This is an 8 item questionnaire, recalling probability of falling asleep in "recent times". The subjects are asked to rate probability of falling asleep in eight different situations. The score for each item ranges from 0 (would never doze) to 3 (high chance of dozing), with the overall score range of 0 to 24. Higher scores represent higher probability of falling asleep.
Time Frame: recorded at the end of run-in month and blinded month
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Verum | Sham
Number analyzed (Participants) | 24 | 27
score on a scale | 0.84 [0.40 to 2.06] | 1.00 [0.17 to 2.28]
Statistical Analysis 1: Comparison: Verum vs Sham; Test type: Superiority or Other; p = 0.83, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.16

12. Secondary Outcome: Epworth Sleepiness Scale Score
Description: Mean difference of Epworth Sleepiness Scale score between run-in month and open label month. The Epworth Sleepiness Scale is used to measure excessive daytime sleepiness. This is an 8 item questionnaire, recalling probability of falling asleep in "recent times". The subjects are asked to rate probability of falling asleep in eight different situations. The score for each item ranges from 0 (would never doze) to 3 (high chance of dozing), with the overall score range of 0 to 24. Higher scores represent higher probability of falling asleep.
Time Frame: Score recorded at the end of run-in and open label month
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Verum | Sham
Number analyzed (Participants) | 24 | 26
score on a scale | 0.50 [-0.85 to 1.85] | 0.35 [-0.59 to 1.28]
Statistical Analysis 1: Comparison: Verum vs Sham; Test type: Superiority or Other; p = 0.92, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.15

ADVERSE EVENTS:
Time Frame: Over the 28 day blinded period, and 28 day open label period for those wishing to continue after completion of the study (total of 8 weeks)
Description: Inquiry regarding adverse events was made at the visits following the blinded and open label period. We also recorded adverse events reported during phone calls with participants during the blinded and open label period.
Groups:
- Verum: Verum : wears active cranial electrostimulation (CES) device for 20 minutes daily for 28 days
- Sham: Sham: wears sham cranial electrostimulation (CES) device for 20 minutes daily for 28 days
Arm/Group | Verum | Sham
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 6/34 | 0/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Verum (N=34) | Sham (N=34)
Visual Flickering (Eye disorders) | 6 (6) | 0 (0) — Sensation of visual flickering related to electrical pulse, was irritating and possibly worsened headache while wearing

LIMITATIONS AND CAVEATS:
Recall bias in completing survey instruments. Incomplete diary data with regards to headache symptoms, acute medication use and relief limited analysis for other proposed secondary outcomes.Higher than anticipated drop-out rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No